CLINICAL TRIAL: NCT06534658
Title: Study on Multimodal Imaging and Molecular Imaging Techniques in Degenerative Dementia
Acronym: MIMI
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BP-MIMI
Record Dates: First submitted 2024-07-18; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease; Image
Keywords: Alzheimer Disease; molecular imaging
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is a multicenter observational study that establishes a longitudinal cohort of patients with Alzheimer's disease and other dementias based on neuroimaging, molecular imaging, biological and digital markers to explore new solutions such as dementia disease mechanism, diagnosis, condition evaluation, and prognosis assessment.

DETAILED DESCRIPTION:
This project will build a longitudinal database based on multimodal MRI imaging information of dementia subjects, various body fluid or digital markers, and a cohort. The convolutional neural network algorithm will be used to explore the imaging characteristics of healthy controls, AD, FTD, and DLB, develop an early prediction model for degenerative dementia, and achieve early differential diagnosis of different dementia subtypes. This study further performed GE180, ASEM, and exendin-4 radionuclide imaging on some subjects who completed conventional PET (AV45, Tauvir, and FDG) imaging to explore the diagnostic efficacy of these three probes as new diagnostic probes for early AD. In addition, through longitudinal follow-up of Aβ-positive MCI patients, multimodal MRI and PET image fusion technology were used to explore the changes in fused images during their conversion to AD in order to obtain early and accurate diagnostic markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥50 and ≤85 years old, male or female;
* Meet the diagnostic criteria for dementia or MCI;
* Neuropsychological score: MMSE 15-28 points, CDR ≤ 1 point; ④ Patients and their families are informed and sign the informed consent form

Exclusion Criteria:

* The presence of other neurological diseases that may cause brain dysfunction (such as depression, brain tumors, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal intracranial pressure hydrocephalus, etc.);
* The presence of other systemic diseases that may cause cognitive impairment (such as liver dysfunction, renal dysfunction, thyroid dysfunction, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.);
* Suffering from a disease that makes it impossible to cooperate with cognitive examinations;
* The presence of contraindications to MRI;
* The presence of mental and neurological retardation;
* Refusing to draw blood;
* Refusing to sign the informed consent form.

Ages: 50 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population in this study includes the cognitive impairment patients in Ruijin Hospital, Renji Hospital, The First Hospital of Zhejiang University School of Medicine, The First Hospital of China Medical University.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2029-07-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
The change of incidence of cognitive impairment | baseline, 1 year, 2 year, 3 year, 4 year
  Number of participants who covert to AD or mild cognitive impairment (MCI) will be recorded to calculate the incidence.

SECONDARY OUTCOMES:
The change of Mini-Mental State Examination (MMSE) | baseline, 1 year, 2 year, 3 year, 4 year
  MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures) in elderly participants. Total score ranges from 0 to 30; lower score indicates greater disease severity.
The change of Montreal cognitive assessment-Basic (MoCA) | baseline, 1 year, 2 year, 3 year, 4 year
  MoCA is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures) in elderly participants. Total score ranges from 0 to 30; lower score indicates greater disease severity.
The change of Auditory verbal learning test (AVLT) | baseline, 1 year, 2 year, 3 year, 4 year
  AVLT is a screening instrument used to assess the function of memory. The score in long-term memory (N5) ranges from 0 to 12, with lower scores indicating greater disease severity.
The change of structural MRI | baseline, 1 year, 2 year, 3 year, 4 year
  Structural MRI data will be acquired and analyzed through high-resolution T1-weighted MRI and diffusion tensor imaging (DTI).
The change of functional MRI | baseline, 1 year, 2 year, 3 year, 4 year
  Functional MRI data will be acquired and analyzed through blood oxygenation level dependent (BOLD) imaging.
The change of magnetic susceptibility | baseline, 1 year, 2 year, 3 year, 4 year
  Magnetic susceptibility data will be acquired and analyzed through quantitative susceptibility mapping (QSM)
The change of perfusion MR imaging | baseline, 1 year, 2 year, 3 year, 4 year
  Perfusion imaging data will be acquired and analyzed through arterial spin labeling (ASL).
Positron emission tomography (PET)-MRI | baseline, 1 year, 2 year, 3 year, 4 year
  Including AV45-PET, FDG-PET, Tau-PET, GLP-1R PET, Cholinergic receptor probe (ASEM) PET will be used to detect the amyloid, Tau burden and AD related GLP-1R as well as Cholinergic receptor change
The change of blood biomarker | baseline, 1 year, 2 year, 3 year, 4 year
  Blood serum p-tau 181, p-tau 217, Aβ40, pEAβ3-42 and Aβ42 , GFAP, NFL at baseline will be tested. The higher blood p-tau is a strong predictor for AD.
The change of speech information | baseline, 1 year, 2 year, 3 year, 4 year
  Voice data collection, use a voice recorder to collect the patient's description of "stealing biscuit map" language, and save it in SWV format. And use self-developed ASR speech analysis software (China software copyright number: 2016RS164680) for speech analysis.
The change of Activities of daily living (ADL) | baseline, 1 year, 2 year, 3 year, 4 year
  ADL is a scale used in healthcare to refer to people's daily self-care activities. Eight factors are rated to produce an overall score on a point scale of 0 to 100. The lower the score the more independence in living.
The change of Geriatric Depression Scale (GDS) | baseline, 1 year, 2 year, 3 year, 4 year
  GDS is a neuropsychological scale used to assess the level of depression. The total score ranges from 0 to 30, with higher scores indicating greater disease severity.
The change of electroencephalogram (EEG) | baseline, 1 year, 2 year, 3 year, 4 year
  Electroencephalogram (EEG) is used to measure electrical activity in the brain using small, metal discs (electrodes) attached to the scalp. Recorded frequencies include alpha, beta, delta and theta band power. The EEG signatures of people with cognitive impairment will be further analyzed, and its longitudinal changes will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, PhD. MD., Principal Investigator — RenJi Hospital
Locations (8):
- China (8):
  - Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hanzhong, Hangzhou
  - Cangzhou Hospital of Integrated Traditional Chinese and Western Medicine, Cangzhou, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Qilu Hospital of Shandong University, Qingdao Branch, Qingdao, Shandong
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of China Medical University, Shenyang, Shenyang